CLINICAL TRIAL: NCT01636141
Title: A Phase 1, Randomized, Dose Escalation, Single Center, Safety Study of Single and Multi-Dose, Topically Applied OLT1177 Gel in Healthy Subjects
Brief Title: Phase 1 Safety Study of Single and Multi-Dose Topically Applied OLT1177 Gel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OLT1177-01
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Pharmacokinetics; Dose escalation; Randomized; Healthy volunteers; Topical; OLT1177; Olatec; Pain; Inflammation
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo gel (Placebo Comparator): Each study group consists of 6 subjects randomized in a 5:1 ratio to receive OLT1177 Gel or placebo gel in both Part A and B of the study. Eighteen subjects will be enrolled in Part A and 18 in Part B. A total of 30 subjects will receive OLT1177 Gel and 6 subjects will receive placebo gel.
  Interventions: Drug: Placebo gel
- OLT1177 Gel (Active Comparator): Each study group consists of 6 subjects randomized in a 5:1 ratio to receive OLT1177 Gel or placebo gel in both Part A and B of the study. Eighteen subjects will be enrolled in Part A and 18 in Part B. A total of 30 subjects will receive OLT1177 Gel and 6 subjects will receive placebo gel.
  Interventions: Drug: OLT1177 Gel

INTERVENTIONS:
Drug: OLT1177 Gel — OLT1177 Gel - 3% or 5% administered topically to a defined area of one knee
  Arms: OLT1177 Gel
Drug: Placebo gel
  Arms: Placebo gel

SUMMARY:
The purpose of this study is to determine if OLT1177 Gel is safe and can be tolerated when given as a single dose and multidose to a defined area of one knee of healthy subjects.

DETAILED DESCRIPTION:
OLT1177 Gel is being developed for the topical treatment of pain and inflammation emanating from musculoskeletal and certain skin inflammatory conditions.

This is a Phase 1 study evaluating the safety and tolerability of OLT1177 Gel in healthy subjects when given as single-dose or multi-dose applications. The study will be conducted in two parts, Part A and Part B. In Part A, approximately 18 healthy subjects in 3 dose escalating cohorts will be randomized to receive a single dose of the investigational drug (5 subjects OLT1177 Gel and 1 subject placebo gel). Upon completion of Part A, a new subject population of approximately 18 subjects in 3 dose escalating cohorts will be randomized in Part B of the study. Subjects will receive a total of 8 doses over 3 consecutive days given 6 hours apart while awake during the day and will be followed for up to 30 days for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 18 to 60 years of age
* Women of childbearing potential must have a negative urine pregnancy test within 3 days of study enrollment and must agree to use a highly effective form of contraception
* Subjects must be in good health as determined by the Investigator based on medical history, ECG, physical examination and safety laboratory test
* Ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the Investigator, to comply with all the requirements of the study

Exclusion Criteria:

* Subjects with a known hypersensitivity to the investigational drug
* Subjects who are pregnant or lactating
* Participation in any investigational drug or device study and receipt of any investigational drug or device within the immediate 30 days prior to the start of this study
* Concurrent or recent use of analgesics, steroids, allergy medications, H2 blockers within 48 hours of the start of the study
* Subjects with a prior knee injury or surgery within the last 5 years
* Subjects with an active infection or with a fever ≥ 38°C within 3 days of the start of the study
* Subjects with a history of, or known to be positive for, HIV, hepatitis B or C
* Subjects with uncontrolled hypertension as defined by systolic blood pressure (SBP) > 150 mm/Hg, diastolic blood pressure (DBP) > 100 mm/Hg
* Subjects with a wound or skin irritation or any skin condition, e.g., psoriasis in the treatment area
* Subjects who are taking prescription medications with the exception of oral or systemic contraceptives
* Subjects who have systemic diseases
* Subjects who have a history of anaphylactic reactions to any systemic or topical compounds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Recording of adverse events | Part A - during the 7 days following the application of the study drug and Part B during the 14 day following each application of the study drug
  Adverse events will be described with respect to seriousness, intensity, relationship to treatment, action taken and outcome of the event.
  Local skin irritation will be assessed at each visit based on individual signs and symptoms of skin tolerability for erythema, pruritus, scaling/dryness, edema and stinging/burning.

SECONDARY OUTCOMES:
Area under the Concentration curve (AUC) | Part A - Pre-dose, 15 minutes, 30 minutes, 1, 2, 4 and 6 hours post dose and Days 2, 3 and 7. Part B - Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, and 6 hours post dose, Days 2, 3 (15 minutes, 30 minutes, 1, 2, 4 and 6 hours post dose) Days 4, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Terry M Jones, MD, Principal Investigator — J&S Studies
Locations (1):
- J&S Studies, Inc, College Station, Texas, United States